CLINICAL TRIAL: NCT03164421
Title: N-Acetylcysteine Versus L-carnitine in Clomiphene Citrate Resistant Pcos Women. a Randomized Controlled Trial
Brief Title: N-Acetylcysteine and L-carnitine in Pcos
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZUH 7
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2017-06

CONDITIONS: PCOS
MeSH Terms: interventions — Acetylcysteine; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-Acetylcysteine (Experimental): N-Acetylcysteine used by clomiphene resistant pcos women
  Interventions: Drug: N-Acetylcysteine
- L-carnitine (Active Comparator): L-carnitine used by clomiphene resistant pcos women
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine in clomiphene resistant pcos women
  Arms: N-Acetylcysteine
Drug: L-carnitine — L-carnitine in clomiphene resistant pcos women
  Other Names: motova plus
  Arms: L-carnitine

SUMMARY:
N-Acetylcysteine and L-carnitine were used in pcos patients

DETAILED DESCRIPTION:
N-Acetylcysteine was compared to L-carnitine in clomiphene citrate in Pcos women to detect the hormonal and metabolic effect

ELIGIBILITY:
Inclusion Criteria:

* pco
* infertile

Exclusion Criteria:

* no medical disorders
* no hormonal treatment in the previous 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 3 momths
  number of women with clinical pregnancy

SECONDARY OUTCOMES:
ovulation rate | 3 momths
  number of women with follicle >18mm.
abortion rate | 3 momths
  number of women with abortions

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A EL sharkwy, MD, Principal Investigator — FACULTY OF MEDICINE ,ZAGAZIG UNIVERSITY
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the collected data willbe available within 6 months

REFERENCES:
- [Derived] El Sharkwy IA, Abd El Aziz WM. Randomized controlled trial of N-acetylcysteine versus l-carnitine among women with clomiphene-citrate-resistant polycystic ovary syndrome. Int J Gynaecol Obstet. 2019 Oct;147(1):59-64. doi: 10.1002/ijgo.12902. Epub 2019 Jul 17. PMID 31273783